CLINICAL TRIAL: NCT01541657
Title: Sensory-Targeted Ankle Rehabilitation Strategies
Brief Title: Sensory-Targeted Ankle Rehabilitation Strategies (STARS)
Acronym: STARS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Joel Thompson (Other)
Collaborators: Ithaca College (Other); University of North Carolina, Charlotte (Other); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor-Investigator, Joel Thompson, UK PRS Adminstrator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R03AR06156101
Record Dates: First submitted 2012-02-20; First posted 2012-03-01 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Chronic Ankle Instability
Keywords: Ankle Instability; Sensorimotor Control; Sensory; Postural Control; Balance; Gait
MeSH Terms: interventions — Pliability

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control Group (No Intervention): This group will only take part in the data collection sessions. After the first testing session (Pre-Intervention) the participants will be asked to rest comfortably for 5 minutes. After the rest period, they will be reassessed. Upon completion of the second testing, they will be asked to maintain the same lifestyle over the course of 2 weeks. They will then be asked to return to the lab after the 2 week interval to be tested again. Upon completion of the third testing session, they will be contacted after 1 month to complete the self-reported function questionnaires.
- Ankle Joint Mobilization (Experimental): The posterior ankle mobilization treatment is a manual therapy technique that consists of gently gliding your ankle in the backward direction through a pain free range of motion. This is a common therapy technique used by athletic trainers for the treatment of ankle sprains. The objective of this therapy technique is to glide the ankle into the area which restricts range of motion and gently stretch the restricted area. To begin this treatment, a certified athletic trainer with experience in applying this therapy technique will provide mild traction to the ankle joint to lightly distract the bones of the ankle joint. The athletic trainer will then apply two sets of joint mobilizations which will each last 2 minutes. Each repetition will consist of gently gliding the ankle joint in the backward direction until an area of restriction is reached. The athletic trainer will push into the restriction and then glide the ankle back to the starting position.
  Interventions: Other: Ankle Joint Mobilization
- Foot Massage (Experimental): The foot massage treatment is a manual therapy technique that consists of gently rubbing the bottom of your feet with both hands like kneading dough. To begin the treatment, you will be asked to lie comfortably on a treatment table you're your feet hanging slightly off the edge. The athletic trainer with experience in applying this therapy will place his hands on the bottom of your foot and begin to massage your feet from your toes down to your heel. The athletic trainer will perform 2 sets of 2 minutes of massage with 1 minute rest in between sets.
  Interventions: Other: Foot Massage
- Calf Stretching (Experimental): The calf stretching treatment is a technique that is commonly used in sports and rehabilitation. You will be asked to place your foot on a slant board located next to a wall with your heel positioned below your toes on the slant board. You will be asked to lean towards the wall until you feel tension in your calf muscles that feels like a good stretch. You will perform 2 sets of 3 stretches that are held for 30 seconds each. Between each stretch, you will rest for 10 seconds. Between each set, you will rest for 1 minute.
  Interventions: Other: Calf Stretching

INTERVENTIONS:
Other: Ankle Joint Mobilization — The posterior ankle mobilization treatment is a manual therapy technique that consists of gently gliding your ankle in the backward direction through a pain free range of motion. This is a common therapy technique used by athletic trainers for the treatment of ankle sprains. The objective of this therapy technique is to glide the ankle into the area which restricts range of motion and gently stretch the restricted area. To begin this treatment, a certified athletic trainer with experience in applying this therapy technique will provide mild traction to the ankle joint to lightly distract the bones of the ankle joint. The athletic trainer will then apply two sets of joint mobilizations which will each last 2 minutes. Each repetition will consist of gently gliding the ankle joint in the backward direction until an area of restriction is reached. The athletic trainer will push into the restriction and then glide the ankle back to the starting position.
  Other Names: Ankle Range of Motion; Joint Manipulation
  Arms: Ankle Joint Mobilization
Other: Foot Massage — The foot massage treatment is a manual therapy technique that consists of gently rubbing the bottom of your feet with both hands like kneading dough. To begin the treatment, you will be asked to lie comfortably on a treatment table you're your feet hanging slightly off the edge. The athletic trainer with experience in applying this therapy will place his hands on the bottom of your foot and begin to massage your feet from your toes down to your heel. The athletic trainer will perform 2 sets of 2 minutes of massage with 1 minute rest in between sets.
  Other Names: Plantar Massage; Plantar Stimulation; Foot Rub
  Arms: Foot Massage
Other: Calf Stretching — The calf stretching treatment is a technique that is commonly used in sports and rehabilitation. You will be asked to place your foot on a slant board located next to a wall with your heel positioned below your toes on the slant board. You will be asked to lean towards the wall until you feel tension in your calf muscles that feels like a good stretch. You will perform 2 sets of 3 stretches that are held for 30 seconds each. Between each stretch, you will rest for 10 seconds. Between each set, you will rest for 1 minute.
  Other Names: Muscle Stretch; Flexibility
  Arms: Calf Stretching

SUMMARY:
The purpose of this study is to determine the effect of 3 types of sensory-targeted rehabilitation interventions on subjective and objective measures of function for those with chronic ankle instability. The investigators hypothesize that subjective and objective measures of function including self-reported disability, balance, and range of motion will improve after 2-weeks of sensory-targeted interventions.

DETAILED DESCRIPTION:
The purpose of this study is to determine the effect of 3 types of sensory-targeted rehabilitation interventions on subjective and objective measures of function for those with chronic ankle instability. If a potential participant is deemed eligible for participation and consents to participate, he/she undergo a pretest session in which balance, gait, and range of motion will be assessed. The participant will then be randomized into one of the 4 treatment groups and undergo the first treatment which takes approximately 5 minutes. After completion of the first treatment, the participant will be immediately retested on the balance, gait, and range of motion measures. Upon completion of testing on the first day, participants in the treatment groups will be asked to return for 5 more treatments over the course of 2 weeks. Upon completion of the treatments, each participant will be tested on their balance, gait, and range of motion again. Then, after 1 month, each participant will be contacted to do a self-reported function follow-up visit in which he/she will be asked to report how stable and functional his/her ankle has been over the past month.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18-45 years of age
2. History of ankle sprain with at least two episodes of "giving way" within the past six months
3. Score of ≥ 5 on the Ankle Instability Instrument (AII)
4. Score of ≤ 90% on the Foot and Ankle Ability Measure (FAAM)- Activity of Daily Living (ADL) Subscale
5. Score of ≤ 80% on the FAAM-Sport Subscale.

Exclusion Criteria:

1. Younger than 18 or older than 45 years
2. No history of ankle sprain or episodes of "giving way" in the past six months
3. Score of ≤ 5 on the Ankle Instability Instrument (AII)
4. Score of ≥ 90% on the FAAM-ADL
5. Score of ≥ 80% on the FAAM-S.
6. An acute ankle sprain within the past 6 weeks.
7. Previous history of lower extremity surgery with internal derangements, reconstructions, or repair
8. Lower extremity injury within the past 6 months (other than ankle sprains)
9. Presence of balance deficits or conditions known to affect balance as noted on the Balance Questionnaire including diabetes and/or vertigo.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2011-12; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Foot and Ankle Ability Measure | This will be assessed at 3 time points: Change from Pre-intervention to Post-Intervention, change from Pre-Intervention to 1-month Post-Intervention
  The Foot and Ankle Ability Measure (FAAM) is a questionnaire used to quantify the amount of self-reported disability a person experiences because of chronic ankle instability. It has two sections which will be used to assess disability associated with activities of daily living and sport activities.
Gait Initiation | This will be assessed at 3 time points: Change from Pre-Intervention to Immediately Post Day 1 Intervention, and Change from Pre-Intervention to Post-Intervention
  Gait initiation is a laboratory technique that involves the use of a force plate. Participants are asked to stand on the force plate with feet and step off the force plate with either the right or left foot. The size of the weight shifts a participant makes while taking a step are evaluated using the force plate. Each participant will complete 5 trials stepping with each leg for every time point.
Time to Boundary | This will be assessed at 3 time points: Change from Pre-Intervention to Immediately Post Day 1 Intervention, and Change from Pre-Intervention to Post-Intervention
  Time to Boundary is a balance measurement in which a person maintains single leg stance on a force plate for 10 seconds. This measurement technique evaluates the amount of time a person has to make corrections to maintain balance. Each participant will perform 12 trials for each time point. Each leg will be tested 6 times, 3 with eyes open and 3 with eyes closed.
Weight-bearing Lunge Test | This will be assessed at 3 time points: Change from Pre-Intervention to Immediately Post Day 1 Intervention, and Change from Pre-Intervention to Post-Intervention
  The Weight-bearing Lunge Test is a measure of ankle dorsiflexion range of motion while the participant stands in front of a wall.
Cutaneous Sensation | This will be assessed at 3 time points: Change from Pre-Intervention to Immediately Post Day 1 Intervention, and Change from Pre-Intervention to Post-Intervention
  Each participant will have the sensitivity of the bottom of his/her feet assessed. The investigators will use a set of monofilaments (similar to fishing line) to see how small of a monofilament can be detected when the investigator touches the bottom of his or her foot. Participants will be asked to close their eyes during testing.
Single Limb Balance Error Scoring System Assessment | This will be assessed at 3 time points: Change from Pre-Intervention to Immediately Post Day 1 Intervention, and Change from Pre-Intervention to Post-Intervention
  Each participant will be asked to balance on one leg for 20 seconds with eyes closed while standing on the floor. During the test, the investigator will count how many times the participant deviates from the target position (standing on one leg with hands on hips).

CONTACTS AND LOCATIONS:
Overall Officials: Patrick O McKeon, PhD, Principal Investigator — Ithaca College; Erik A Wikstrom, PhD, Principal Investigator — University of North Carolina, Charlotte
Locations (2):
- United States (2):
  - Ithaca College, Ithaca, New York
  - University of North Carolina Charlotte, Charlotte, North Carolina

REFERENCES:
- [Derived] McKeon PO, Wikstrom EA. The effect of sensory-targeted ankle rehabilitation strategies on single-leg center of pressure elements in those with chronic ankle instability: A randomized clinical trial. J Sci Med Sport. 2019 Mar;22(3):288-293. doi: 10.1016/j.jsams.2018.08.017. Epub 2018 Sep 6. PMID 30244979